CLINICAL TRIAL: NCT04197817
Title: A Randomized, Double-blind, Placebo-controlled, Single-dose Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of JS002 (Recombinant Humanized Anti-PCSK9 Monoclonal Antibody) Injection in Healthy Subjects.
Brief Title: A Single Dose Escalation Study of PCSK9 Inhibitor (JS002) in Health Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: JS002-001
Record Dates: First submitted 2019-12-01; First posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JS002 (Active Comparator): JS002, Subcutaneous or intravenous injection
  Interventions: Drug: JS002
- Placebo, (Placebo Comparator): Placebo,Subcutaneous or intravenous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JS002 — JS002, Subcutaneous or intravenous injection of a single dose of JS002, dose cohort according to ascending dose design
  Other Names: Recombinant humanized Anti- PCSK9 monoclonal antibody
  Arms: JS002
Drug: Placebo — Placebo,Subcutaneous or intravenous injection of a single dose of placebo, dose cohort according to ascending dose design
  Other Names: Placebo of Recombinant humanized Anti- PCSK9 monoclonal antibody
  Arms: Placebo,

SUMMARY:
JS002 is a recombinant humanized Anti- PCSK9 monoclonal antibody; This is a phase Ia, randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of a single subcutaneous injection of JS002 in healthy subjects.

In this study, the dose ascending design includes five dose level cohorts (15 mg, 50 mg, 150 mg, 300 mg, and 450 mg) administered by subcutaneous injection, and three intravenous administration cohorts (15 mg, 150 mg, and 450 mg). Each cohort will enroll 8 to 12 subjects (distribution of study drug and placebo in a 3:1 ratio).

The duration of the study is 84-day per subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men or women aged 18 to 45 years old at screening visit;
2. Have the ability to read and understand, volunteer to participate in the study, and signed written informed consent.
3. The body mass index (BMI) at screening visit was in the range of 18 to 30 kg/m2 (inclusive) and the body weight ≥ 50 kg.
4. The sitting blood pressure ≥90/60 mmHg and <140/90 mmHg at screening visit.
5. Serum LDL-C level ≥ 70 mg/dL (1.8 mmol/L) and < 190 mg/dL (4.9 mmol/L) at screening visit.
6. Serum Triglyceride (TG) level < 250 mg/dL (2.8 mmol/L) at screening visit.
7. No fertility [female: documented hysterectomy, bilateral oophorectomy, tubal ligation or other female permanent sterilization, or menopause (menopause for more than one year)], or those with fertility are willing to take, during the entire study period, strict and effective contraceptive measures, in addition, female subjects with fertility should have a negative blood/urine pregnancy test at screening visit.

Exclusion Criteria:

1. Subjects who meet any of the following criteria will be excluded from the study:
2. Evolocumab and/or Alirocumab, or other targeted drugs to PCSK9, has been used at any time.
3. Any therapeutic or research biological agents has been used during the first 6 months of baseline/random (Day 0).
4. Participated in any clinical study within 3 months prior to baseline/random (Day 0).
5. Any drug or health supplement that affects blood lipids or lipid metabolism during the first 30 days of baseline/random (Day 0), including but not limited to: Probucol, statins (e.g. Atorvastatin, Rosuvastatin, etc.), cholesterol absorption inhibitors (such as Ezetimibe), bile acid sequestrants (such as Cholestyramine), red yeast and hawthorn preparations, fibrates, high-purity fish oil preparations (or omega-fatty acids ≥ 1000 mg / day) and niacin preparation (nicotinic acid ≥ 50 mg), etc.
6. Start a new intense exercise or diet control within 30 days of random (Day 0) or major changes to previous diet and lifestyle (including exercise, smoking and drinking). The following conditions occur before the baseline/random (Day 0) 1 day (ie Day-1) need to be excluded:

   * Creatine kinase (CK) ≥ 3 times the upper limit of normal (ULN) (Note: related to exercise), or
   * Urinary cotinine is positive, or
   * Positive alcohol saliva test.
7. Previous or concomitant diseases (such as nephrotic syndrome, liver disease, diabetes, hypothyroidism, etc.) or any clinically significant abnormalities found in physical examinations, laboratory tests, and electrocardiograms, which would make the subject unsuitable for this study.
8. The medical history or clinical evidence indicates that the subject had severe acute or chronic disease (including not limited to: heart, kidney, nerves, endocrine, blood, immunity, infection, metabolic disorders, etc.), and the disease has not been controlled, which may confuse the outcome of the study or put the subject at risk judged by the investigator, The following situations need to be excluded:

   * had major surgery in the last 6 months, or
   * has been hospitalized (e.g. infection) in the last 3 months, or
   * donated blood or blood loss ≥500 mL in the past 3 months, or
   * has used any prescription or over-the-counter drugs in the past 1 month.
9. Transplantation History of organs (such as heart, lung, liver, kidney, etc.) Malignant tumors history, except for cervical carcinoma in situ or surgically resected skin cancer (basal cells and squamous epithelial cells) for more than 5 years.
10. Drug abuse or alcohol dependence in the past 1 year.
11. HIV infection, or HIV antibody positive at screening visit.
12. Syphilis infection, or serotonin antibody (TPPA) positive at screening visit.
13. Hepatitis B surface antigen (HBsAg) was positive at screening visit.
14. Hepatitis C virus (HCV) antibody was positive at screening visit.
15. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≥ 2 times the upper limit of normal (ULN); alkaline phosphatase and bilirubin ≥ 1.5 times the upper limit of normal (ULN).
16. Allergy history to mammalian-derived biological agents, including monoclonal antibodies.
17. Women during pregnancy and lactation.
18. Any other investigator believes that the subject is not suitable for the study, such as the subject has potential compliance issues, cannot complete all tests and assessments according to the protocol requirements.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2018-08-14 (Actual); Study Completion 2018-08-14 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events（SAE, drug-related (S)AE etc）based on physical examinations, vital signs, 12 lead ECGs , laboratory tests and injection site reactions. | Up to 84 days after dose administration

SECONDARY OUTCOMES:
Number of participants with anti-drug antibodies. | Up to 84 days after dose administration
Serum concentrations of JS002 at different timepoint after the drug administration. | Up to 84 days after dose administration
Change from baseline in LDL-C and other lipid parameters (TC, HDL-C, non-HDL-C, VLDL-C, ApoB, ApoA1, Lp(a) and TG). | Up to 84 days after dose administration

OTHER OUTCOMES:
Changes over time of serum concentrations of JS002. | Up to 84 days after dose administration
Changes over time of LDL-C. | Up to 84 days after dose administration
Change over time of unbound/total serum PCSK9. | Up to 84 days after dose administration

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China